CLINICAL TRIAL: NCT00123591
Title: A Randomised, Double-Blind, Placebo-Controlled, Multi-centre, Dose Escalation Study to Evaluate the Safety and Preliminary Efficacy of Recombinant Factor VIIa (NovoSeven®/NiaStase®) in Subjects With Brain Contusions
Brief Title: Safety and Preliminary Efficacy of Recombinant Activated Factor VII in Subjects With Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7CBI-1600; 2004-000088-92 (EudraCT Number)
Record Dates: First submitted 2005-06-30; First posted 2005-07-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Asia, Europe, Middle East, and North America. The primary objective of the trial is to evaluate the safety of Recombinant Activated Factor VII in patients with brain contusions. The secondary objective of the trial is to evaluate the preliminary efficacy of Recombinant Activated Factor VII in preventing early haemorrhagic progression in contusive brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Contusive brain injury (including brain stem) diagnosed by history, clinical examination and confirmed by CT scan within 6 hours of onset
* In British Columbia and Nova Scotia, subjects must be = 19 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the Safety of Recombinant Activated Factor VII in Subjects with Brain Contusions | Within the first 15 days of injury

SECONDARY OUTCOMES:
Evaluate the preliminary efficacy of Recombinant Activated Factor VII in preventing haemorrhagic progression in brain contusions

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- Novo Nordisk Investigational Site, Montreal, Canada
- Novo Nordisk Investigational Site, Helsinki, Finland
- Novo Nordisk Investigational Site, Hanover, Germany
- India (2):
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Bangalore
- Israel (3):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Ramat Gan
  - Novo Nordisk Investigational Site, Tel Aviv
- Novo Nordisk Investigational Site, Cesena, Italy
- Novo Nordisk Investigational Site, Rotterdam, Netherlands
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Barcelona, Spain
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Taoyuan District, Taiwan

REFERENCES:
- [Result] Narayan RK, Maas AI, Marshall LF, Servadei F, Skolnick BE, Tillinger MN; rFVIIa Traumatic ICH Study Group. Recombinant factor VIIA in traumatic intracerebral hemorrhage: results of a dose-escalation clinical trial. Neurosurgery. 2008 Apr;62(4):776-86; discussion 786-8. doi: 10.1227/01.neu.0000316898.78371.74. PMID 18496183
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com